CLINICAL TRIAL: NCT06161857
Title: Auditory Brainstem Response Thresholds at 6 and 8KHz in Adults With Normal Hearing and Sensorineural Hearing Loss
Brief Title: High Frequency ABR
Status: Recruiting | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: 8537; 32889 (Other: IRAS)
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hearing Loss, High-Frequency
MeSH Terms: conditions — Hearing Loss, High-Frequency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Hearing Group: Participants with hearing levels of 20dBHL or better at 6 and 8kHz frequencies of sound
  Interventions: Other: No intervention
- Mild Hearing Loss Group: Participants with hearing levels of 25-40dBHL at 6 and 8kHz frequencies of sound
  Interventions: Other: No intervention
- Moderate Hearing Loss Group: Participants with hearing levels of 45-70dBHL at 6 and 8kHz frequencies of sound
  Interventions: Other: No intervention
- Severe Hearing Loss Group: Participants with hearing levels of 75- 90dBHL at 6 and 8kHz frequencies of sound
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention this is an observational study to develop a diagnostic test

SUMMARY:
This study is looking at a method called 'ABR', which measures the electrical activity in the brain (brain waves) when we hear sounds. This study will look at the electrical activity in participants brains in response to high-pitched sounds. First, the investigators will find the quietest sounds the participants can hear. Then the investigators will use 'ABR' to measure the quietest sounds that trigger electrical activity in participants brains'. This is to find out if there is a difference between the quietest sounds participants can hear, and the quietest sounds that trigger these brain waves. We are also interested in finding out if having a hearing loss affects this.

DETAILED DESCRIPTION:
The most common way of measuring how good someone's hearing is, is to play them sounds at different levels and ask them to respond when they can hear it, for example, by pressing a button when they hear a sound. However, some people such as young children and people with learning disabilities can't do this. So, we may use the ABR technique instead. However, there are usually differences between ABR thresholds (the quietest level of sound needed to trigger an electrical response in the brain) and behavioural hearing level thresholds (the quietest level sound is perceived). If we know what this difference usually is, we can use ABR to work out how good someone's hearing is. We can already do this for most of the important pitches (aka frequencies) of sound, as typically experienced in the muffled sound in telephones. But we do not know the difference between ABR and behavioural thresholds for high-pitched sounds that help make hearing crisper. So, that is what this study is trying to find out.

To do this we need people with different hearing levels to participate in our study. Including people with normal hearing and people with a hearing loss. We aim to recruit nearly 40 people in total with a range of different hearing levels.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able and willing to give informed consent.
* Participant is over 18.
* Hearing in the test ear of ≤90dBSPL at 6 kHz and 8 kHz in PTA
* Able and willing to perform PTA reliably.
* Able and willing to sit still comfortably for the duration of an ABR.

Exclusion Criteria:

* Any conductive element to hearing loss (air-bone gap on PTA of >10dB).
* Occluding wax, TM perforations or ear infections (on otoscopy)
* CI or BAHA user
* Abnormal outer of middle ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study needs a range of participants with different hearing levels.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Difference between ABR and PTA thresholds | through study completion, 4-5 months
  Compare ABR thresholds to PTA thresholds at 6 and 8 kHz in normal hearing adults and adults with sensorineural hearing loss.

SECONDARY OUTCOMES:
Effect of participants hearing level on ABR-PTA threshold differences | through study completion, 4-5 months
  Analyse the effect of hearing level on ABR-PTA threshold differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and Value University Health Board, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No